CLINICAL TRIAL: NCT04746313
Title: Assessment of the Prevalence of Hyperprolactinemia in Systemic Scleroderma
Brief Title: Prevalence of Hyperprolactinemia in Systemic Scleroderma
Acronym: SCLERO-PRL
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Association pour la Formation et la Recherche en Médecine Interne (AFORMI) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020_18; 2020-A03066-33 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2021-02-08; First posted 2021-02-09 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Sclerosis, Systemic; Scleroderma; Hyperprolactinemia
Keywords: Systemic sclerosis; Scleroderma; Prolactin
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Hyperprolactinemia | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with systemic sclerosis: The study will be systematically offered to any scleroderma patient seen in scheduled hospitalization
  Interventions: Biological: blood test
- Healthy subjects: Healthy subjects who will donate blood to the French Blood Establishment (EFS) and matched to scleroderma patients on age (+/- 5 years) and sex
  Interventions: Biological: blood test

INTERVENTIONS:
Biological: blood test — * to analysis prolactin in healthy subjects and scleroderma patients
  * then to analysis in only scleroderma patients: thyroid-stimulating hormone (TSH), thyroxine (T4), luteinizing hormone (LH), oestradiol, follicle-stimulating hormone (FSH), BAFF (B-cell activating factor), IL-6 (interleukin 6) and endoglin

SUMMARY:
Systemic sclerosis is an autoimmune and inflammatory disease characterized primarily by fibrosis and vascular involvement. We know that the immune system is disrupted in systemic sclerosis, but there are probably other mechanisms to explain the disease, including deregulation of certain proteins such as prolactin

ELIGIBILITY:
Inclusion Criteria:

Scleroderma patients:

* man or woman over 18 years old
* with systemic sclerosis meeting ACR-EULAR 2013 criteria
* having given his no opposition
* being social insured

Healthy subjects:

* man or woman over 18 years old
* donation of blood to the EFS
* matched on age (+/- 5 years) and sex
* having given his no opposition

Exclusion Criteria:

* Man or woman under 18 years old
* Pregnant or breastfeeding women
* Receiving medical treatment inducing dysfunction of the hypothalamic pituitary axis
* Refusing or unable to give no objection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Scleroderma patients are from scheduled hospitalization Department of Internal Medicine and Clinical Immunology, CHU Lille Healthy subjects are from the French Blood Establishment (EFS) and matched to scleroderma patients on age (+/- 5 years) and sex
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
the prevalence of hyperprolactinemia in scleroderma patients | At 2 years
  Rate of prolactin measured by immuno-chemiluminescence (Abbott Architect automaton).
  The presence of a defined hyperprolactinemia at the University Hospital of Lille: for women, prolactin level higher than 26.5 ng/mL and for men, higher than 19.4 ng/mL.

SECONDARY OUTCOMES:
the prevalence of hyperprolactinemia between scleroderma patients and healthy subjects matched by age and sex | At 2 years
the associations between prolactin levels and clinical (scleroderma phenotype, visceral involvement) and biological (inflammation, antibodies, cytokines) manifestations in systemic sclerosis | At 2 years
association between prolactin levels and biological markers of the immune system in scleroderma patients | At 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David Launay, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France

IPD SHARING:
Plan to Share IPD: Undecided